CLINICAL TRIAL: NCT00730691
Title: A Randomized, Double-Blind, Parallel-Group, Placebo-Controlled, Active-Referenced, Fixed-Dose Study Comparing the Efficacy and Safety of 3 Doses of Lu AA21004 in Acute Treatment of Adults With Generalized Anxiety Disorder
Brief Title: Efficacy of Vortioxetine (Lu AA21004) in Treating Generalized Anxiety Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LuAA21004_308; U1111-1114-3966 (Registry Identifier: WHO)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Mood Disorder; Affective Disorder; Anxiety Disorder; Drug Therapy
MeSH Terms: conditions — Generalized Anxiety Disorder; Mood Disorders; Anxiety Disorders | interventions — Vortioxetine; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo-matching capsules, orally, once daily for up to 9 weeks.
  Interventions: Drug: Placebo
- Vortioxetine 2.5 mg (Experimental): Vortioxetine 2.5 mg encapsulated tablets, orally, once daily, for 8 weeks, followed by placebo-matching capsules, orally, once daily, for 1 week.
  Interventions: Drug: Placebo; Drug: Vortioxetine
- Vortioxetine 5 mg (Experimental): Vortioxetine 5 mg encapsulated tablets, orally, once daily, for 8 weeks, followed by placebo-matching capsules, orally, once daily, for 1 week.
  Interventions: Drug: Placebo; Drug: Vortioxetine
- Vortioxetine 10 mg (Experimental): Vortioxetine 10 mg encapsulated tablets, orally, once daily, for 8 weeks, followed by placebo-matching capsules, orally, once daily, for 1 week.
  Interventions: Drug: Placebo; Drug: Vortioxetine
- Duloxetine 60 mg (Active Comparator): Duloxetine 60 mg capsules, orally, once daily, for 8 weeks, followed by duloxetine 30 mg capsules, orally, once daily, for 1 week.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Placebo — Placebo-matching capsules
  Arms: Placebo; Vortioxetine 10 mg; Vortioxetine 2.5 mg; Vortioxetine 5 mg
Drug: Vortioxetine — Encapsulated vortioxetine immediate release tablets
  Other Names: Lu AA21004; Brintellix®
  Arms: Vortioxetine 10 mg; Vortioxetine 2.5 mg; Vortioxetine 5 mg
Drug: Duloxetine — Overencapsulated duloxetine capsules
  Other Names: Cymbalta
  Arms: Duloxetine 60 mg

SUMMARY:
The purpose of this study is to determine the safety and efficacy of vortioxetine, once daily (QD), in adults with generalized anxiety disorder.

DETAILED DESCRIPTION:
Participants in this study will be randomly assigned to receive either 2.5 mg, 5 mg or 10 mg of vortioxetine, once daily, 60 mg of duloxetine once daily, or a placebo once daily for eight weeks.

Participants will be seen weekly during the first 2 weeks of treatment, and then every 2 weeks up to the end of the 8-week treatment period. Participants who complete the 8-week treatment period will enter a 2-week discontinuation period in order to assess potential discontinuation symptoms. Total commitment time is up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has a primary diagnosis of generalized anxiety disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR®) criteria (classification code 300.02).
* Has a Hamilton Anxiety Scale total score ≥ 20. Has a Hamilton Anxiety Scale score ≥2 on both item 1 (anxious mood) and item 2 (tension).
* Has a Montgomery-Åsberg Depression Rating Scale total score ≤16.

Exclusion Criteria:

* Had received any investigational compound <30 days before Screening or 5 half-lives prior to Screening, whichever is longer.
* Received Lu AA21004 in a previous clinical study.
* Was a study site employee, or an immediate family member (ie, spouse, parent, child, or sibling) of a study site employee involved in conduct of this study.
* Has 1 or more of the following:

  * Any current psychiatric disorder other than Generalized Anxiety Disorder as defined in the DSM-IV-TR® (as assessed by the Mini International Neuropsychiatric Interview [MINI]).
  * Current or past history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including major depression with psychotic features, mental retardation, organic mental disorders, or mental disorders due to a general medical condition as defined in the DSM-IV-TR.
  * Any substance disorder (except nicotine and caffeine) within the previous 6 months as defined in the DSM-IV-TR® and must have a negative urine drug screen prior to Baseline.
  * Presence or history of a clinically significant neurological disorder (including epilepsy).
  * Neurodegenerative disorder (Alzheimer disease, Parkinson disease, multiple sclerosis, Huntington disease, etc).
  * Any Axis II disorder that might compromise the study.
* Has known sensitivity to duloxetine.
* Is taking excluded medications
* Has a significant risk of suicide according to the investigator's opinion or has a score ≥5 on item 10 (suicidal thoughts) of the Montgomery-Åsberg Depression Rating Scale or has made a suicide attempt in the previous 6 months.
* Has previously failed to respond to adequate treatment with selective serotonin reuptake inhibitor and/or serotonin-norepinephrine reuptake inhibitors.
* Has received electroconvulsive therapy within 6 months prior to Screening.
* Is currently receiving formal cognitive or behavioral therapy, systematic psychotherapy, or plans to initiate such therapy during the study.
* Has a known history of or currently has increased intraocular pressure or is at risk of acute narrow-angle glaucoma.
* Has a clinically significant unstable illness, for example, hepatic impairment or renal insufficiency, or a cardiovascular, pulmonary, gastrointestinal, endocrine, neurological, rheumatologic, immunologic, infectious, skin and subcutaneous tissue disorders, or metabolic disturbance.
* Has an alanine aminotransferase, aspartate aminotransferase, or total bilirubin level >1.5 times the upper limit of normal.
* Has a serum creatinine level >1.5 upper limit of normal.
* Has a previous history of cancer that had been in remission for less than 5 years.
* Hasclinically significant abnormal vital signs as determined by the investigator.
* Has a history of lack of response to previous adequate treatment with duloxetine for any Generalized Anxiety Disorder episode.
* Has 1 or more laboratory values outside the normal range, based on the blood or urine samples taken at the Screening Visit
* Has a thyroid stimulating hormone value outside the normal range.
* Has an abnormal electrocardiogram.
* has a disease or was taking medications that, in the opinion of the investigator, could have interfered with the assessments of safety, tolerability, or efficacy.
* The patient, in the opinion of the investigator, was unlikely to comply with the clinical study protocol or was unsuitable for any reason.
* Had previously been enrolled in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 781 (Actual)
Dates: Start 2008-06; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (66):
- United States (66):
  - Anaheim, California
  - Beverly Hills, California
  - Fresno, California
  - Los Angeles, California
  - Oceanside, California
  - San Diego, California
  - Sherman Oaks, California
  - Widomar, California
  - Denver, Colorado
  - Farmington, Connecticut
  - Norwalk, Connecticut
  - Coral Gables, Florida
  - Jacksonville, Florida
  - Maitland, Florida
  - Miami, Florida
  - Orlando, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - Winter Park, Florida
  - Atlanta, Georgia
  - Roswell, Georgia
  - Smyrna, Georgia
  - Honolulu, Hawaii
  - Oakbrook Ter, Illinois
  - Terre Haute, Indiana
  - Owensboro, Kentucky
  - Shreveport, Louisiana
  - Rockville, Maryland
  - Chesterfield, Missouri
  - St Louis, Missouri
  - Nashua, New Hampshire
  - Clementon, New Jersey
  - Princeton, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Cedarhurst, New York
  - New York, New York
  - Rochester, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Beachwood, Ohio
  - Cleveland, Ohio
  - Dayton, Ohio
  - Toledo, Ohio
  - Eugene, Oregon
  - Portland, Oregon
  - Salem, Oregon
  - Allentown, Pennsylvania
  - Media, Pennsylvania
  - Philadelphia, Pennsylvania
  - Columbia, South Carolina
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - DeSoto, Texas
  - Houston, Texas
  - Lake Jackson, Texas
  - Wichita Falls, Texas
  - Midvale, Utah
  - Woodstock, Vermont
  - Richmond, Virginia
  - Seattle, Washington
  - Brown Deer, Wisconsin
  - Middleton, Wisconsin
  - Milwaukee, Wisconsin

REFERENCES:
- [Derived] Mahableshwarkar AR, Jacobsen PL, Chen Y, Simon JS. A randomised, double-blind, placebo-controlled, duloxetine-referenced study of the efficacy and tolerability of vortioxetine in the acute treatment of adults with generalised anxiety disorder. Int J Clin Pract. 2014 Jan;68(1):49-59. doi: 10.1111/ijcp.12328. PMID 24341301

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 71 investigative sites in the United States from 20 June 2008 to 27 February 2009.
Pre-assignment Details: Participants with a diagnosis of generalized anxiety disorder were enrolled equally in 1 of 5 treatment groups, once a day placebo, 2.5 mg, 5 mg or 10 mg vortioxetine, or 60 mg duloxetine.
Groups:
- Vortioxetine 5 mg: Vortioxetine 5 mg encapsulated tablets, orally, once daily, for 8 weeks, followed by placebo-matching capsule, orally, once daily, for 1 week.
Period: Overall Study
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Started | 157 | 156 | 156 (One participant was randomized by error. Reason not completed is reported as Other.) | 156 | 156
Completed | 121 | 120 | 117 | 111 | 106
Not Completed | 36 | 36 | 39 | 45 | 50
Not completed — Adverse Event | 4 | 8 | 11 | 11 | 23
Not completed — Lack of Efficacy | 4 | 4 | 2 | 1 | 1
Not completed — Non-compliance with Study Drug | 6 | 1 | 6 | 3 | 3
Not completed — Protocol Deviations | 3 | 5 | 3 | 7 | 5
Not completed — Withdrawal of Consent | 7 | 9 | 3 | 6 | 3
Not completed — Lost to Follow-up | 11 | 8 | 13 | 15 | 13
Not completed — Other | 1 | 1 | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg | Total
Number analyzed (Participants) | 157 | 156 | 156 | 156 | 156 | 781
Age Continuous [Mean (Standard Deviation); unit: years] | 36.8 (12.12) | 39.2 (11.90) | 37.7 (11.96) | 39.8 (12.33) | 39.5 (12.28) | 38.6 (12.14)
Age, Customized [Number; unit: participants]
  ≤55 years | 143 | 140 | 147 | 137 | 137 | 704
  >55 years | 14 | 16 | 9 | 19 | 19 | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 109 | 100 | 105 | 113 | 529
  Male | 55 | 47 | 56 | 51 | 43 | 252
Race/Ethnicity, Customized [Number; unit: participants] — Race data only available for 154 participants in the vortioxetine 2.5 mg arm.
  participants
    Caucasian (White, including Hispanic) | 118 | 121 | 124 | 120 | 121 | 604
    Black | 35 | 31 | 26 | 33 | 31 | 156
    Asian | 4 | 0 | 6 | 0 | 4 | 14
    American Indian or Alaska Native | 0 | 1 | 0 | 2 | 0 | 3
    Native Hawaiian/ Other Pacific Islander | 0 | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 157 | 156 | 156 | 156 | 156 | 781
Weight [Mean (Standard Deviation); unit: kg] | 84.40 (25.426) | 79.47 (19.893) | 80.98 (20.312) | 80.17 (21.420) | 79.51 (20.090) | 80.91 (21.558)
Height [Mean (Standard Deviation); unit: cm] | 168.74 (9.605) | 167.87 (9.139) | 169.25 (9.282) | 167.61 (8.378) | 167.94 (9.300) | 168.28 (9.147)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.54 (8.478) | 28.19 (6.651) | 28.24 (6.589) | 28.49 (7.058) | 28.10 (6.325) | 28.51 (7.064)
Smoking Classification [Number; unit: participants] — Smoking classification data available for 156 participants in the placebo arm.
  participants
    Never Smoked | 92 | 85 | 81 | 85 | 82 | 425
    Current Smoker | 41 | 43 | 44 | 43 | 43 | 214
    Ex-smoker | 23 | 28 | 31 | 28 | 31 | 141
Alcohol Consumption [Number; unit: participants] — Alcohol consumption data available for 156 participants in the placebo arm.
  participants
    Never | 40 | 49 | 40 | 53 | 44 | 226
    Once monthly or less often | 71 | 50 | 66 | 49 | 64 | 300
    Once a week | 27 | 25 | 31 | 29 | 19 | 131
    2 to 6 times per week | 17 | 30 | 17 | 22 | 22 | 108
    Daily | 1 | 2 | 2 | 3 | 7 | 15
Hamilton Anxiety Scale Total Score [Mean (Standard Deviation); unit: scores on a scale] — Hamilton Anxiety Scale (HAM-A) is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (absent) to 56 (maximum severity).
  scores on a scale | 24.4 (3.73) | 25.3 (4.25) | 25.0 (3.57) | 25.3 (3.96) | 25.0 (3.94) | 25.0 (3.90)
Clinical Global Impression - Severity scale score [Mean (Standard Deviation); unit: scores on a scale] — The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale where the clinician rates the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
  scores on a scale | 4.3 (0.56) | 4.4 (0.63) | 4.4 (0.59) | 4.4 (0.59) | 4.4 (0.62) | 4.4 (0.60)
Hospital Anxiety and Depression - Anxiety subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Anxiety sub-scale consists of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). The anxiety subscale determines a state of generalized anxiety including anxious mood, restlessness, anxious thoughts and panic attacks. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 13.9 (3.23) | 13.8 (3.40) | 13.8 (3.70) | 14.0 (3.02) | 13.4 (3.70) | 13.8 (3.41)
Hospital Anxiety and Depression - Depression subscale [Mean (Standard Deviation); unit: scores on a scale] — Hospital Anxiety and Depression (HAD) Depression sub-scale consists of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). The depression subscale focuses on the state of lost interest and diminished pleasure response. Scores are summed and range from 0 to 21 (maximal severity).
  scores on a scale | 8.2 (4.12) | 8.2 (3.83) | 8.2 (3.94) | 8.5 (3.59) | 8.2 (4.00) | 8.2 (3.89)
Montgomery Åsberg Depression Rating Scale (MADRS) total score [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery Åsberg Depression Rating Scale (MADRS) is a depression rating scale consisting of 10 items, each rated 0 to 6. The 10 items represent the core symptoms of depressive illness. The overall score ranges from 0 (symptoms absent) to 60 (severe depression).
  scores on a scale | 11.83 (2.787) | 12.24 (3.279) | 12.24 (2.895) | 12.47 (2.868) | 11.99 (3.087) | 12.16 (2.989)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Anxiety (HAM-A) Scale Total Score at Week 8
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. Least Squares (LS) means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Week 8
Population: The full analysis set (FAS) included all randomized patients who received at least 1 dose of study drug, and had at least 1 postbaseline value for assessment of primary efficacy. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 120 | 118 | 114 | 111 | 106
scores on a scale | -11.27 (0.595) | -12.23 (0.600) | -11.57 (0.606) | -11.66 (0.606) | -13.87 (0.635)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; P-values were tested at the 5% level of significance (ie, statistical significance if P<0.05) comparing each of the 3 doses of vortioxetine to placebo; Test type: Superiority or Other; p = 0.255, Mixed model for repeated measurements — This treatment arm is not in the pre-specified testing sequence, a nominal p-value is provided; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.96, 95% CI 2-sided [-2.62 to 0.69], Standard Error of Mean 0.843
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; To control for multiplicity, a pre-specified sequential testing procedure was applied to compare 10 mg and 5 mg vortioxetine to placebo; as soon as an endpoint was non-significant at 0.025, the testing procedure stopped for all subsequent endpoints; Test type: Superiority or Other; p = 0.719, Mixed model for repeated measurements — Pre-specified sequential statistical testing procedure indicates that when p-value >0.025, hierarchical testing stops and for subsequent endpoints in the sequence a nominal p-value is provided; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.30, 95% CI 2-sided [-1.96 to 1.35], Standard Error of Mean 0.843
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.642, Mixed model for repeated measurements — [p-value comment as in outcome 1, analysis 2]; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.39, 95% CI 2-sided [-2.06 to 1.27], Standard Error of Mean 0.848
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.003, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -2.60, 95% CI 2-sided [-4.30 to -0.89], Standard Error of Mean 0.869

2. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HAD) - Anxiety Subscale at Week 8
Description: The HAD-Anxiety subscale is completed by the participant and measures anxiety, including anxious mood, restlessness, anxious thoughts, and panic attacks. The subscale is made up of 7 items that are assessed on a scale from 0 (no anxiety) to 3 (severe feeling of anxiety). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. Scores are summed and range from 0 to 21 (maximal severity). LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 123 | 120 | 119 | 111 | 108
scores on a scale | -4.00 (0.361) | -3.89 (0.364) | -4.24 (0.366) | -5.09 (0.372) | -5.54 (0.385)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.830, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = 0.11, 95% CI 2-sided [-0.89 to 1.11], Standard Error of Mean 0.511
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.643, Mixed model for repeated measurements — Hierarchical testing stopped at the primary endpoint in the testing sequence, a nominal p-value is provided; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.24, 95% CI 2-sided [-1.24 to 0.77], Standard Error of Mean 0.510
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.036, Mixed model for repeated measurements — Hierarchical testing stopped at the primary endpoint in the testing sequence, a nominal p-value is provided; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -1.09, 95% CI 2-sided [-2.10 to -0.07], Standard Error of Mean 0.517
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.004, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS mean Difference = -1.54, 95% CI 2-sided [-2.58 to -0.50], Standard Error of Mean 0.527

3. Secondary Outcome: Mean Clinical Global Impression Scale-Global Improvement (CGI-I) at Week 8
Description: The Clinical Global Impression - Global Improvement scale measures the participant's improvement (or worsening) as assessed by the investigator relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 120 | 118 | 114 | 111 | 106
scores on a scale | 2.47 (0.091) | 2.36 (0.092) | 2.38 (0.093) | 2.38 (0.093) | 2.03 (0.098)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.407, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.11, 95% CI 2-sided [-0.36 to 0.15], Standard Error of Mean 0.129
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.533, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.08, 95% CI 2-sided [-0.33 to 0.17], Standard Error of Mean 0.129
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.491, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.09, 95% CI 2-sided [-0.34 to 0.17], Standard Error of Mean 0.130
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.001, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.44, 95% CI 2-sided [-0.70 to -0.17], Standard Error of Mean 0.133

4. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Week 8
Description: The Sheehan Disability Scale assesses functional impairment in 3 domains: work/school, social life or leisure activities, and home life or family responsibilities. The participant rates the extent to which each aspect is impaired on a 10-point visual analog scale, from 0 (not at all) to 10 (extremely). The 3 scores are added together to calculate the total score, which ranges from 0 to 30, with higher scores indicating more impairment. LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Week 8
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 97 | 94 | 95 | 94 | 84
scores on a scale | -6.35 (0.631) | -6.15 (0.647) | -6.68 (0.642) | -7.95 (0.623) | -8.81 (0.675)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.652, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = 0.35, 95% CI 2-sided [-1.16 to 1.85], Standard Error of Mean 0.765
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.511, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.50, 95% CI 2-sided [-1.98 to 0.98], Standard Error of Mean 0.754
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.204, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -0.94, 95% CI 2-sided [-2.38 to 0.51], Standard Error of Mean 0.736
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.001, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -2.57, 95% CI 2-sided [-4.10 to -1.03], Standard Error of Mean 0.781

5. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Week 8
Description: Response was defined as participants with a ≥50% decrease from Baseline in the HAM-A total score. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Week 8
Population: Full analysis set; Last observation carried forward (LOCF) was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 149
percentage of participants | 42.2 | 44.8 | 42.6 | 44.8 | 51.0
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.641, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 1.114, 95% CI 2-sided [0.709 to 1.750]
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.945, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 1.016, 95% CI 2-sided [0.643 to 1.605]
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.641, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 1.114, 95% CI 2-sided [0.709 to 1.749]
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.124, Regression, Logistic; Logistic regression with explanatory variables for treatment and Baseline HAM-A score; Odds Ratio (OR) = 1.427, 95% CI 2-sided [0.907 to 2.246]

6. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Week 8 in Participants With Baseline HAM-A ≥25
Description: The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 to 56 where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe. Total scores above 30 are rare, but indicate very severe anxiety. LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Week 8
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 52 | 60 | 60 | 50 | 48
scores on a scale | -11.61 (1.008) | -14.12 (0.945) | -13.87 (0.955) | -13.22 (0.999) | -16.15 (1.039)
Statistical Analysis 1: Comparison: Placebo vs Vortioxetine 2.5 mg; Test type: Superiority or Other; p = 0.064, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -2.50, 95% CI 2-sided [-5.15 to 0.14], Standard Error of Mean 1.346
Statistical Analysis 2: Comparison: Placebo vs Vortioxetine 5 mg; Test type: Superiority or Other; p = 0.096, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -2.26, 95% CI 2-sided [-4.92 to 0.40], Standard Error of Mean 1.353
Statistical Analysis 3: Comparison: Placebo vs Vortioxetine 10 mg; Test type: Superiority or Other; p = 0.250, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -1.61, 95% CI 2-sided [-4.36 to 1.14], Standard Error of Mean 1.397
Statistical Analysis 4: Comparison: Placebo vs Duloxetine 60 mg; Test type: Superiority or Other; p = 0.002, Mixed model for repeated measurements; P-values are from an MMRM model with week, Baseline score-by-week and treatment-by-week interaction as factors; LS Mean Difference = -4.54, 95% CI 2-sided [-7.34 to -1.73], Standard Error of Mean 1.425

7. Secondary Outcome: Change From Baseline in Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed
Description: as for outcome 6
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: Full analysis set. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 149
scores on a scale
  Week 1 (n= 151, 149, 142, 149, 143) | -4.70 (0.423) | -4.56 (0.421) | -4.90 (0.430) | -5.04 (0.419) | -5.48 (0.435)
  Week 2 (n=147, 145, 143, 147, 130) | -7.30 (0.472) | -7.28 (0.471) | -8.22 (0.476) | -7.63 (0.468) | -9.29 (0.494)
  Week 4 (n= 139, 135, 132, 133, 116) | -8.66 (0.518) | -9.77 (0.520) | -9.84 (0.525) | -9.73 (0.519) | -11.13 (0.553)
  Week 6 (n= 127, 123, 122, 120, 112) | -10.28 (0.547) | -10.82 (0.553) | -11.26 (0.556) | -11.05 (0.552) | -12.66 (0.583)

8. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HAD) - Anxiety Subscale at Other Weeks Assessed
Description: as for outcome 2
Time Frame: Baseline to Weeks 1 and 4
Population: Full analysis set with available data at Baseline. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 148
scores on a scale
  Week 1 (n=150, 149, 141, 149, 141) | -1.81 (0.273) | -1.85 (0.274) | -1.89 (0.280) | -2.22 (0.272) | -2.91 (0.285)
  Week 4 (n=141, 142, 139, 141, 126) | -3.24 (0.310) | -3.34 (0.310) | -3.60 (0.313) | -4.01 (0.310) | -5.11 (0.328)

9. Secondary Outcome: Mean Clinical Global Impression Scale-Global Improvement (CGI-I) at Other Weeks Assessed
Description: The Clinical Global Impression - Global Improvement scale measures the participant's improvement (or worsening) as assessed by the clinician relative to Baseline on a 7-point scale: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse. LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Weeks 1, 2, 4 and 6
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 147 | 154 | 148
scores on a scale
  Week 1 (n=151, 148, 141, 149, 141) | 3.44 (0.067) | 3.46 (0.068) | 3.41 (0.069) | 3.40 (0.067) | 3.36 (0.070)
  Week 2 (n=147, 145, 142, 147, 129) | 3.03 (0.072) | 3.08 (0.072) | 2.90 (0.073) | 2.96 (0.072) | 2.76 (0.077)
  Week 4 (n=140, 135, 132, 134, 116) | 2.81 (0.079) | 2.67 (0.080) | 2.67 (0.081) | 2.68 (0.080) | 2.44 (0.085)
  Week 6 (n=127, 123, 121, 120, 112) | 2.61 (0.082) | 2.53 (0.083) | 2.43 (0.084) | 2.41 (0.083) | 2.25 (0.088)

10. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) at Other Weeks Assessed
Description: as for outcome 4
Time Frame: Baseline to Weeks 1, 2 and 4
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 126 | 121 | 118 | 133 | 119
scores on a scale
  Week 1 (n=116, 111, 109, 125, 112) | -3.22 (0.506) | -2.74 (0.521) | -3.28 (0.521) | -4.11 (0.483) | -4.74 (0.521)
  Week 2 (n=116, 114, 116, 123, 103) | -4.53 (0.536) | -4.18 (0.547) | -5.02 (0.542) | -5.46 (0.514) | -7.09 (0.563)
  Week 4 (n=108, 106, 106, 115, 91) | -4.55 (0.590) | -4.98 (0.604) | -5.92 (0.600) | -6.47 (0.568) | -7.95 (0.632)

11. Secondary Outcome: Percentage of Responders in HAM-A Total Score at Other Weeks Assessed
Description: as for outcome 5
Time Frame: Baseline and Weeks 1, 2, 4 and 6
Population: Full analysis set; LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 149
percentage of participants
  Week 1 (n=151, 149, 142, 149, 143) | 11.3 | 6.7 | 8.5 | 10.1 | 16.8
  Week 2 (n=154, 154, 147, 154, 149) | 20.8 | 20.1 | 21.1 | 21.4 | 28.9
  Week 4 (n=154, 154, 148, 154, 149) | 26.0 | 30.5 | 32.4 | 35.1 | 42.3
  Week 6 (n=154, 154, 148, 154, 149) | 36.4 | 37.7 | 40.5 | 40.9 | 47.7

12. Secondary Outcome: Change From Baseline in the Hamilton Anxiety Scale (HAM-A) Total Score at Other Weeks Assessed in Participants With Baseline HAM-A ≥25
Description: as for outcome 6
Time Frame: Baseline to weeks 1, 2, 4 and 6
Population: Full analysis set patients with a HAM-A Baseline score ≥25. A mixed model for repeated measurements (MMRM) based on observed cases was used; "n" indicates the number of patients included in the analysis at each time point.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 65 | 80 | 74 | 73 | 70
scores on a scale
  Week 1 (n=63, 76, 70, 70, 66) | -5.32 (0.787) | -6.07 (0.719) | -5.96 (0.749) | -5.94 (0.740) | -6.78 (0.770)
  Week 2 (n=62, 73, 70, 68, 62) | -7.55 (0.856) | -8.82 (0.785) | -10.18 (0.810) | -8.51 (0.808) | -10.40 (0.844)
  Week 4 (n=60, 68, 67, 63, 54) | -8.61 (0.901) | -11.61 (0.837) | -12.87 (0.854) | -10.98 (0.862) | -12.56 (0.914)
  Week 6 (n=58, 63, 62, 54, 51) | -10.72 (0.937) | -12.86 (0.880) | -14.11 (0.895) | -12.75 (0.918) | -14.35 (0.961)

13. Secondary Outcome: Percentage of Participants in HAM-A Remission at Each Week Assessed
Description: Remission is defined as a Hamilton Anxiety Scale (HAM-A) total score ≤ 7. The HAM-A is an anxiety rating scale consisting of 14 items that assess anxious mood, tension, fear, insomnia, intellectual (cognitive) symptoms, depressed mood, behavior at interview, somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic and somatic (muscular) symptoms. Each symptom is rated from 0 (absent) to 4 (maximum severity). Total scores range from 0 (symptoms absent) to 56 (maximum severity).
Time Frame: Weeks 1, 2, 4, 6 and 8
Population: Full analysis set. LOCF was used. "n" indicates the number of patients included in the analysis at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 149
percentage of participants
  Week 1 (n=151, 149, 142, 149, 143) | 4.0 | 2.0 | 0.7 | 2.0 | 4.9
  Week 2 (n=154, 154, 147, 154, 149) | 6.5 | 8.4 | 7.5 | 3.9 | 12.1
  Week 4 (n=154, 154, 148, 154, 149) | 10.4 | 13.6 | 11.5 | 13.0 | 17.4
  Week 6 (n=154, 154, 148, 154, 149) | 16.2 | 14.9 | 14.9 | 16.9 | 20.8
  Week 8 (n=154, 154, 148, 154, 149) | 22.1 | 20.1 | 19.6 | 20.1 | 28.2

14. Secondary Outcome: Change From Baseline in Clinical Global Impression Scale-Severity of Illness (CGI-S)
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness on the following scale: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill. LS means were from a mixed model for repeated measurements (MMRM) with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Weeks 1, 2, 4, 6 and 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 147 | 154 | 148
scores on a scale
  Week 1 (n=151, 148, 141, 149, 142) | -0.42 (0.055) | -0.37 (0.055) | -0.39 (0.056) | -0.42 (0.054) | -0.54 (0.057)
  Week 2 (n=147, 145, 142, 147, 130) | -0.71 (0.066) | -0.74 (0.066) | -0.80 (0.067) | -0.75 (0.065) | -0.97 (0.069)
  Week 4 (n=140, 135, 132, 134, 115) | -0.95 (0.076) | -1.12 (0.077) | -1.02 (0.077) | -1.11 (0.076) | -1.28 (0.082)
  Week 6 (n=127, 123, 121, 120, 112) | -1.22 (0.083) | -1.32 (0.084) | -1.31 (0.084) | -1.35 (0.084) | -1.55 (0.088)
  Week 8 (n=120, 118, 114, 111, 106) | -1.42 (0.095) | -1.50 (0.096) | -1.38 (0.097) | -1.44 (0.097) | -1.77 (0.101)

15. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression (HAD) - Depression Subscale at All Weeks Assessed
Description: The HAD-Depression subscale is completed by the participant and measures depression, focusing on the state of lost interest and diminished pleasure response. The subscale is made up of 7 items that are assessed on a scale from 0 (no depression) to 3 (severe feeling of depression). Participants are required to indicate the response which most accurately reflects the way they have felt over the last few days. The item scores are summed and the total subscore ranges from 0 to 21 (maximal severity). LS means were from a mixed model for repeated measurements (MMRM) model with week, Baseline score-by-week and treatment-by-week interaction as factors.
Time Frame: Baseline to Weeks 1, 4 and 8
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 148
scores on a scale
  Week 1 (n=150, 149, 141, 149, 141) | -0.81 (0.226) | -0.83 (0.226) | -0.88 (0.231) | -1.25 (0.225) | -1.19 (0.235)
  Week 4 (n=141, 142, 139, 141, 126) | -1.32 (0.268) | -1.83 (0.268) | -1.70 (0.271) | -1.61 (0.268) | -2.62 (0.283)
  Week 8 (n=123, 120, 119, 111, 108) | -2.21 (0.300) | -1.82 (0.303) | -1.96 (0.305) | -1.94 (0.310) | -2.77 (0.320)

16. Secondary Outcome: Health Care Resource Utilization Assessed by the Health Economic Assessment Questionnaire
Description: Healthcare resource utilization was assessed by the Health Economic Assessment (HEA) questionnaire, which monitors the participants absenteeism from work, as well as resource use such as visits to a general practitioner, outpatient and inpatient services, hospitalization, medications, and other relevant services over the past 8 weeks.
Time Frame: Baseline and Week 8
Population: Full analysis set
Measure: Number; unit: participants
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Number analyzed (Participants) | 154 | 154 | 148 | 154 | 149
participants
  Baseline: Any resource use | 34 | 36 | 26 | 43 | 38
  Baseline: Any hospitalization-related services | 0 | 3 | 1 | 0 | 2
  Baseline: Hospitalization related to anxiety | 0 | 2 | 1 | 0 | 0
  Baseline: Any sick leave | 14 | 16 | 13 | 15 | 12
  Baseline: Sick leave related to anxiety | 5 | 10 | 9 | 9 | 7
  Week 8: Any resource use | 26 | 24 | 29 | 23 | 22
  Week 8: Any hospitalization-related service | 0 | 0 | 0 | 1 | 3
  Week 8: Hospitalization related to anxiety | 0 | 0 | 0 | 0 | 1
  Week 8: Any sick leave | 13 | 6 | 7 | 7 | 11
  Week 8: Sick leave related to anxiety | 2 | 2 | 3 | 1 | 4

ADVERSE EVENTS:
Time Frame: From the first dose of double-blind study medication through 30 days after permanent discontinuation of double-blind study medication.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Vortioxetine 2.5 mg | Vortioxetine 5 mg | Vortioxetine 10 mg | Duloxetine 60 mg
Serious Adverse Events (participants affected / at risk) | 0/155 | 1/156 | 0/155 | 1/156 | 3/154
Other Adverse Events (participants affected / at risk) | 85/155 | 100/156 | 104/155 | 111/156 | 116/154
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Vortioxetine 2.5 mg (N=156) | Vortioxetine 5 mg (N=155) | Vortioxetine 10 mg (N=156) | Duloxetine 60 mg (N=154)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
Sexual abuse (Social circumstances) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=155) | Vortioxetine 2.5 mg (N=156) | Vortioxetine 5 mg (N=155) | Vortioxetine 10 mg (N=156) | Duloxetine 60 mg (N=154)
Vision blurred (Eye disorders) | 6 | 2 | 1 | 4 | 4
Nausea (Gastrointestinal disorders) | 27 | 26 | 45 | 53 | 57
Dry mouth (Gastrointestinal disorders) | 10 | 14 | 17 | 21 | 25
Diarrhoea (Gastrointestinal disorders) | 9 | 9 | 11 | 20 | 6
Constipation (Gastrointestinal disorders) | 6 | 10 | 4 | 12 | 8
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 11 | 11 | 3
Vomiting (Gastrointestinal disorders) | 6 | 5 | 5 | 9 | 10
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 2 | 2 | 2
Stomach discomfort (Gastrointestinal disorders) | 1 | 1 | 4 | 1 | 2
Flatulence (Gastrointestinal disorders) | 3 | 4 | 3 | 4 | 1
Fatigue (General disorders) | 3 | 6 | 8 | 9 | 15
Irritability (General disorders) | 4 | 6 | 4 | 4 | 1
Asthenia (General disorders) | 5 | 3 | 0 | 0 | 2
Feeling jittery (General disorders) | 2 | 0 | 1 | 4 | 4
Nasopharyngitis (Infections and infestations) | 7 | 14 | 7 | 12 | 3
Upper respiratory tract infection (Infections and infestations) | 9 | 12 | 11 | 12 | 8
Influenza (Infections and infestations) | 1 | 1 | 6 | 2 | 2
Viral upper respiratory tract infection (Infections and infestations) | 3 | 5 | 6 | 2 | 2
Gastroenteritis (Infections and infestations) | 4 | 1 | 0 | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 4 | 3 | 1 | 1 | 2
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 4 | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 3 | 2 | 5 | 5 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 4 | 2 | 1
Headache (Nervous system disorders) | 20 | 18 | 20 | 25 | 26
Somnolence (Nervous system disorders) | 6 | 7 | 13 | 8 | 18
Dizziness (Nervous system disorders) | 5 | 13 | 9 | 14 | 17
Tension headache (Nervous system disorders) | 1 | 4 | 4 | 5 | 2
Libido decreased (Psychiatric disorders) | 1 | 3 | 7 | 3 | 7
Anorgasmia (Psychiatric disorders) | 0 | 1 | 1 | 2 | 6
Insomnia (Psychiatric disorders) | 4 | 6 | 6 | 5 | 6
Anxiety (Psychiatric disorders) | 2 | 2 | 3 | 2 | 5
Abnormal dreams (Psychiatric disorders) | 0 | 3 | 5 | 2 | 4
Restlessness (Psychiatric disorders) | 2 | 2 | 1 | 5 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2 | 3 | 2 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.